CLINICAL TRIAL: NCT02418871
Title: Clinical Evaluation of the FluidVision Accommodating Intraocular Lens With an Improved Injector System
Brief Title: Evaluation of the FluidVision Accommodating Intraocular Lens (AIOL) With an Improved Injector System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PowerVision (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: AIOL-2015-1
Record Dates: First submitted 2015-04-09; First posted 2015-04-16 (Estimated); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Aphakia
Keywords: Cataract
MeSH Terms: conditions — Aphakia; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- FluidVision (Experimental): FluidVision AIOL implanted in the capsular bag of the eye during cataract surgery
  Interventions: Device: FluidVision AIOL; Procedure: Cataract surgery

INTERVENTIONS:
Device: FluidVision AIOL — Investigational implantable medical device intended for long-term use over the lifetime of the cataract subject. An improved injector system was used.
Procedure: Cataract surgery — Performed using standard microsurgical techniques

SUMMARY:
The purpose of this study is to evaluate the clinical outcomes of an investigational IOL in patients undergoing cataract extraction and intraocular lens implantation using an improved injector system.

ELIGIBILITY:
Key Inclusion Criteria:

* Eligible for primary intraocular lens implantation for the correction of aphakia following cataract extraction;
* Best corrected distance visual acuity worse than 20/40 either with or without a glare source present (e.g. Brightness Acuity Tester);
* Less than or equal to 1.0 diopter (D) of preoperative keratometric astigmatism;
* Willing and able to comply with schedule for follow-up visits for 36 months after surgery.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Systemic disease that could increase the operative risk or confound the outcome (e.g. autoimmune disease, diabetes);
* Taking systemic medications that may confound the outcome or increase the risk to the subject;
* Ocular conditions that may predispose for future complications;
* Previous intraocular or corneal surgery that might confound the outcome of the investigation or increase the risk to the subject;
* Pregnant, lactating during the course of the investigation, or with another condition associated with fluctuation of hormones that could lead to refractive changes;
* Diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal disorders) that are predicted to cause future best corrected visual acuity loss worse than 20/40.
* Other protocol-defined exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-03-13 (Actual); Primary Completion 2016-03-16 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Accommodative amplitude | Month 6
  Accommodative amplitude is a measure of the ability of the eye to focus from a target that is at distance into a target that is near.
Best corrected distance visual acuity (BCDVA) | Month 6
  Visual acuity of the eye will be tested with the correction in place.
Rates of adverse events | Up to Month 36
  Adverse events will be collected from time of enrollment to study exit.

CONTACTS AND LOCATIONS:
Locations (5):
- PowerVision Investigative Site, Budapest, Hungary
- South Africa (4):
  - PowerVision Investigative Site, Claremont, Cape Town
  - PowerVision Investigative Site, Northcliff, Johannesburg
  - PowerVision Investigative Site, Queenswood, Pretoria
  - PowerVision Investigative Site, Somerset West

IPD SHARING:
Plan to Share IPD: No